CLINICAL TRIAL: NCT02138786
Title: A Phase 2 Study of the Safety and Anti-tumor Activity of the Oral Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330) in Patients With Initial or Refractory and/or Relapsed Richter's Transformation (RT)
Brief Title: Selinexor in Initial or Refractory and/or Relapsed Richter's Transformation
Acronym: SIRRT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy at time of interim analysis
Sponsor: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KCP-330-010
Record Dates: First submitted 2014-05-13; First posted 2014-05-15 (Estimated); Results first posted 2020-02-11 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Richter's Transformation
Keywords: Richter's Transformation; Richter's Syndrome; Karyopharm; selinexor; KPT-330; SIRRT; CLL
MeSH Terms: interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- selinexor (Experimental): oral tablets
  * 10 mg & 25 mg (bottled); or
  * 20 mg (blister pack)
  Interventions: Drug: selinexor

INTERVENTIONS:
Drug: selinexor — * 60 mg dose twice weekly, on Days 1 and 3 of weeks 1-4 of each 4-week cycle; dose may be increased to 80 mg after Cycle 1 unless clinically contraindicated (Protocol V.5.0).
  * 60 mg dose twice weekly on Days 1 and 3 of weeks 1-3 of each 4-week cycle; dose may be increased to 80 mg at Cycle 3 Day 1 unless clinically contraindicated (Protocol V.4.0).
  * 60 mg/m² dose, based on BSA, twice weekly, on Days 1 and 3 of weeks 1-3 of each 4-week cycle (Protocol V. 3.0).
  * 60 mg/m² dose, based on BSA, twice weekly, on Days 1 and 3 of weeks 1-4 of each 4-week cycle (Protocol V. < 3.0).
  Other Names: KPT-330

SUMMARY:
This is a multi-center, phase 2, single arm, open-label study of oral selinexor monotherapy in patients with Richter's Transformation, arising in the setting of prior chronic lymphocytic leukemia (CLL), after at least one chemo-immunotherapy regimen for CLL.

DETAILED DESCRIPTION:
Multi-center, phase 2, single arm, open-label study of oral selinexor monotherapy in patients with Richter's Transformation, arising in the setting of prior CLL, documented by histologically confirmed lymphoma, including diffuse large B-cell (DLBCL) and immunoblastic variants. Eligible patients must have had at least one prior regimen for CLL. Approximately 50 patients are anticipated to be treated in this study. Eligible patients following screening will receive selinexor orally twice weekly at a dose of 60 mg. The selinexor dose may be increased to 80 mg after Cycle 1 unless clinically contraindicated. Patients may continue in multiple treatment cycles at a given dose; there is no maximum treatment duration. Each cycle is 28 days. Dose adjustments will be made as appropriate by the investigator.

Patients who were treated twice weekly for weeks 1-3 under a previous version of the protocol may, at the discretion of the investigator, have had the frequency of selinexor dosing increased to twice weekly for weeks 1-4. If there was no contraindicated toxicity, the selinexor dose may have been increased to 80 mg at Cycle 3.

ELIGIBILITY:
Inclusion Criteria:

* Richter's Transformation, arising in the setting of prior CLL, documented by histologically confirmed lymphoma, including large B-cell and immunoblastic variants.
* All patients must have received at least one prior regimen for CLL, including cytotoxic chemotherapy, anti-CD20 monoclonal antibodies, a BTK inhibitor, or a PI3K inhibitor. Patients may have received high dose chemotherapy/autologous stem cell transplant (HDT/ASCT) or allogeneic hematopoietic stem cell transplant (allo SCT).
* One or more measurable (> 1.5 cm in longest dimension) disease sites on CT (preferably PET/CT) or, if CT is contraindicated, MRI (preferably PET/MRI) scans.
* Objective documented evidence of disease progression at study entry
* Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2

Exclusion Criteria:

* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤ 2 weeks prior to Cycle 1 Day 1, except ibrutinib which may be continued until one day prior to initiation of selinexor; radio-immunotherapy 4 weeks prior to Cycle 1 Day 1. Patients must have recovered to Grade ≤ 1 from clinically significant adverse effects.
* Prolymphocytic transformation
* Less than 1 month since completion of autologous stem cell transplantation or less than 3 months since completion of allogeneic stem cell transplantation
* Major surgery within 4 weeks of C1D1
* Impairment of GI function or GI disease that could interfere with the absorption of selinexor, including obstructed GI tract and uncontrolled vomiting or diarrhea.
* Inability or unwillingness to take supportive medications including a centrally acting appetite stimulant (e.g., mirtazapine or olanzapine) and a peripherally acting appetite stimulant (e.g., low dose glucocorticoids or megesterol acetate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (7):
  - University of Arizona Cancer Center, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California-Los Angeles, Santa Monica, California
  - Winship Cancer Institute / Emory University, Atlanta, Georgia
  - Weill Cornell Medical College, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
- Germany (2):
  - University of Ulm, Ulm, Baden-Wurttemberg
  - University Hospital of Cologne, Cologne
- Poland (3):
  - Malopolskie Centrum Medyczne, Krakow
  - Copernicus Memorial Hospital, Department of Hematology, Lodz
  - Maria Skłodowska-Curie Institue of Oncology, Warsaw
- Spain (3):
  - Instituto Clinico Navarra, Pamplona, Pamplona, Navarre
  - Institut Català d'Oncologia Av., Barcelona
  - Hospital Vall Hebron, Barcelona
- United Kingdom (2):
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Churchill Hospital: Cancer and Haematology Centre, Oxford

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study was conducted at 30 clinical investigative sites in the United States and Europe. Of the 30 investigative sites, 15 sites enrolled a total of 27 patients in the study.
  * Date first patient enrolled: 14 November 2014
  * Date last patient completed: 31 August 2016
Pre-assignment Details: Of the 35 total patients screened, 8 patients were screen-failures. Of the 27 enrolled patients, one patient withdrew from the study prior to receiving treatment. Therefore, a total of 26 patients comprised the Safety population.
Groups:
- Selinexor 60 mg/m² (8 Doses/Cycle): 60 mg/m² dose twice weekly for weeks 1-4
- Selinexor 60 mg (6 Doses/Cycle): 60 mg oral dose twice weekly for weeks 1-3
- Selinexor 60 mg (8 Doses/Cycle): 60 mg oral dose twice weekly for weeks 1-4
Period: Overall Study
Arm/Group | Selinexor 60 mg/m² (8 Doses/Cycle) | Selinexor 60 mg (6 Doses/Cycle) | Selinexor 60 mg (8 Doses/Cycle)
Started | 3 | 15 | 8
Completed | 0 | 0 | 0
Not Completed | 3 | 15 | 8
Not completed — Adverse Event | 0 | 2 | 1
Not completed — Death | 1 | 7 | 2
Not completed — Disease Progression | 1 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Patient's Wish | 0 | 2 | 0
Not completed — Sponsor Terminated Study | 0 | 1 | 1
Not completed — Non-Compliance | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population, consisting of all patients who received any amount of study medication.
Groups:
- Selinexor 60 mg/m² (8 Doses/Cycle): 60 mg/m² oral dose twice weekly for Weeks 1-4
- Total: Total of all reporting groups
Arm/Group | Selinexor 60 mg/m² (8 Doses/Cycle) | Selinexor 60 mg (6 Doses/Cycle) | Selinexor 60 mg (8 Doses/Cycle) | Total
Number analyzed (Participants) | 3 | 15 | 8 | 26
Age, Continuous [Median (Full Range); unit: years] | 68.0 [66 to 74] | 68.0 [41 to 77] | 69.0 [65 to 79] | 68.0 [41 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 4 | 9
  Male | 1 | 12 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 1 | 14 | 8 | 23
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 15 | 8 | 26
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
ECOG score [Count of Participants; unit: Participants] — Performance Status as measured by Eastern Cooperative Oncology Group (ECOG) Status Scale:
  Score=0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction.
  Score=1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  Score=2: In bed < 50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    Score=0 | 0 | 5 | 2 | 7
    Score=1 | 3 | 6 | 4 | 13
    Score=2 | 0 | 4 | 1 | 5
    Missing | 0 | 0 | 1 | 1
Weight [Median (Full Range); unit: kg] — kilograms
  kg | 56.5 [52.3 to 96.0] | 76.5 [51.9 to 115.5] | 73.05 [46.4 to 88.1] | 74.40 [46.4 to 115.5]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Response (Overall Response Rate)
Description: Overall Response Rate (ORR) is defined as the point estimate of the percentage of patients who have complete response (CR) or partial response (PR). Disease response was assessed using the International Working Group (IWG) Response Criteria for non-Hodgkin's lymphoma (Cheson 2007), including assessment of lymph node, spleen and liver lesions by PET (positron emission tomography) scan and assessment of bone marrow biopsies by morphologic, immunohistochemistry, and flow cytometry tests. CR was defined as disappearance of all evidence of disease, and PR was defined as ≥ 50% regression of measurable disease and no new sites.
Time Frame: Assessments were performed at Screening or Cycle 1/Day 1 prior to dosing and on Cycle 3/Day 1 and alternate cycles thereafter until disease progression, study drug intolerability had been reached, study withdrawal, or death.
Population: Modified Intent to Treat (mITT) population, consisting of all patients who received at least one dose of selinexor and had at least one post-baseline efficacy evaluation. Patients without post-baseline efficacy follow-up information who discontinued the study due to toxicity, disease progression, or death were included in this population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Selinexor: All dosing groups
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Percentage of participants | 4 [0.1 to 20.4]

2. Primary Outcome: Number of Participants With Complete Response (CR)
Description: Number of patients who achieved CR (complete disappearance of all detectable evidence of disease). Disease response was assessed using the International Working Group (IWG) Response Criteria for non-Hodgkin's lymphoma (Cheson 2007), including assessment of lymph node, spleen and liver lesions by PET (positron emission tomography) scan and assessment of bone marrow biopsies by morphologic, immunohistochemistry, and flow cytometry tests.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Participants | 0

3. Primary Outcome: Number of Participants With Partial Response (PR)
Description: Number of patients whose best overall response to study treatment was PR (≥ 50% regression of measurable disease and no new sites). Disease response was assessed using the International Working Group (IWG) Response Criteria for non-Hodgkin's lymphoma (Cheson 2007), including assessment of lymph node, spleen and liver lesions by PET (positron emission tomography) scan and assessment of bone marrow biopsies by morphologic, immunohistochemistry, and flow cytometry tests.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Participants | 1

4. Primary Outcome: Number of Participants With Stable Disease (SD)
Description: Number of patients whose best overall response to study treatment was SD (failure to attain criteria for CR or PR, or to meet criteria for PD). Disease response was assessed using the International Working Group (IWG) Response Criteria for non-Hodgkin's lymphoma (Cheson 2007), including assessment of lymph node, spleen and liver lesions by PET (positron emission tomography) scan and assessment of bone marrow biopsies by morphologic, immunohistochemistry, and flow cytometry tests.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Participants | 6

5. Primary Outcome: Number of Participants With Progressive Disease (PD)
Description: Number of patients whose best overall response to study treatment was PD (any new lesion or increase by ≥ 50% of previously involved sites from nadir). Disease response was assessed using the International Working Group (IWG) Response Criteria for non-Hodgkin's lymphoma (Cheson 2007), including assessment of lymph node, spleen and liver lesions by PET (positron emission tomography) scan and assessment of bone marrow biopsies by morphologic, immunohistochemistry, and flow cytometry tests.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Participants | 7

6. Primary Outcome: Number of Participants With Not Evaluable (NE) Response
Description: Number of patients who could not be assessed quantitatively for disease response for any reason.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Participants | 11

7. Secondary Outcome: Percentage of Participants With Disease Control (Disease Control Rate)
Description: Disease Control Rate (DCR) is defined as the percentage of patients who achieved CR, PR, or SD lasting for at least 8 weeks. CR was defined as disappearance of all evidence of disease. PR was defined as ≥ 50% regression of measurable disease and no new sites. SD was defined as failure to attain criteria for CR or PR, or to meet criteria for PD. Disease response was assessed using the International Working Group (IWG) Response Criteria for non-Hodgkin's lymphoma (Cheson 2007), including assessment of lymph node, spleen and liver lesions by PET (positron emission tomography) scan and assessment of bone marrow biopsies by morphologic, immunohistochemistry, and flow cytometry tests.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Percentage of participants | 28.0 [12.1 to 49.4]

8. Secondary Outcome: Duration of Progression Free Survival (PFS)
Description: Number of days calculated from date of start of study therapy to date of progression based on IWG criteria, or date of death if progression did not occur. Patients who dropped out prior to study end without evidence of disease progression were censored at the day they were last known to be alive. Patients without documented disease progression or recurrence were censored at the date of last disease assessment. Disease response was assessed using the International Working Group (IWG) Response Criteria for non-Hodgkin's lymphoma (Cheson 2007), including assessment of lymph node, spleen and liver lesions by PET (positron emission tomography) scan and assessment of bone marrow biopsies by morphologic, immunohistochemistry, and flow cytometry tests.
  .
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Selinexor
Number analyzed (Participants) | 25
Days | 38.0 [22.0 to 86.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected from the first day of dosing (Cycle 1 Day 1) through the 30-day follow-up.
Arm/Group | Selinexor 60 mg/m² (8 Doses/Cycle) | Selinexor 60 mg (6 Doses/Cycle) | Selinexor 60 mg (8 Doses/Cycle)
All-Cause Mortality (participants affected / at risk) | 1/3 | 8/15 | 2/8
Serious Adverse Events (participants affected / at risk) | 3/3 | 9/15 | 5/8
Other Adverse Events (participants affected / at risk) | 3/3 | 15/15 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor 60 mg/m² (8 Doses/Cycle) (N=3) | Selinexor 60 mg (6 Doses/Cycle) (N=15) | Selinexor 60 mg (8 Doses/Cycle) (N=8)
Sepsis (Infections and infestations) | 0 | 1 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
General Physical Health Deterioration (General disorders) | 0 | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Food Intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1
Embolism Arterial (Vascular disorders) | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0
Clostridium Test Positive (Investigations) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Selinexor 60 mg/m² (8 Doses/Cycle) (N=3) | Selinexor 60 mg (6 Doses/Cycle) (N=15) | Selinexor 60 mg (8 Doses/Cycle) (N=8)
Nausea (Gastrointestinal disorders) | 2 | 8 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 5 | 3
Vomiting (Gastrointestinal disorders) | 1 | 7 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 0
Anal Incontinence (Gastrointestinal disorders) | 0 | 2 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Tongue Coated (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 6 | 2
Fatigue (General disorders) | 2 | 4 | 2
Asthenia (General disorders) | 1 | 4 | 2
Oedema Peripheral (General disorders) | 0 | 5 | 1
General Physical Health Deterioration (General disorders) | 1 | 1 | 0
Mucosal Inflammation (General disorders) | 1 | 1 | 0
Early Satiety (General disorders) | 0 | 0 | 1
Facial Pain (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 8 | 5
Anaemia (Blood and lymphatic system disorders) | 1 | 5 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 2 | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 1 | 1
Oral Infection (Infections and infestations) | 0 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 1
Bacteriuria (Infections and infestations) | 0 | 0 | 1
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 1
Device Related Infection (Infections and infestations) | 0 | 1 | 0
Herpes Ophthalmic (Infections and infestations) | 0 | 1 | 0
Oral Herpes (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 4
Headache (Nervous system disorders) | 0 | 3 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1 | 0
Horner's Syndrome (Nervous system disorders) | 0 | 1 | 0
Hypokinesia (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Migraine With Aura (Nervous system disorders) | 0 | 1 | 0
Nervous System Disorder (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Visual Field Defect (Nervous system disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 2
Haematoma (Vascular disorders) | 1 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1
Hot Flush (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Pallor (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0
Post Procedural Contusion (Vascular disorders) | 0 | 1 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 2 | 1
Weight Decreased (Investigations) | 0 | 0 | 3
C-Reactive Protein Increased (Investigations) | 0 | 2 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 2 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0
Blood Creatinine Phophokinase Decreased (Investigations) | 0 | 1 | 0
Blood Creatinine Phosphokinase Increased (Investigations) | 1 | 0 | 0
Hypophonesis (Investigations) | 0 | 1 | 0
International Normalised Ratio Increased (Investigations) | 0 | 1 | 0
Protein Total Decreased (Investigations) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 0 | 1
Eye Irritation (Eye disorders) | 0 | 1 | 0
Ocular Toxicity (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skain Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Tumour Associated Fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Oedema Genital (Reproductive system and breast disorders) | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The low number of formal objective responses (leading to the termination of the study following the first stage), coupled with the high number of censored observations, limited meaningful analyses and the ability to draw conclusions from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes